CLINICAL TRIAL: NCT04325126
Title: Retinol-binding Protein 4 (RBP4) Metabolizm in Type 2 Diabetes Progression and Associated Cardiovascular Complications
Acronym: RMTACC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU 2020 G-66
Record Dates: First submitted 2020-03-26; First posted 2020-03-27 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A total of 500 Chinese patients admitted to the First Affliated Hospital of Xi'an Jiaotong University (Xi'an, China) between March 2020 and March 2022 were recruited to investigate the RBP4 profles. Peripheral blood samples were drawn at the initial medical examination, in the morning after a fast of at least 8 h, and immediately stored at -80˚C until the sphingolipid measurements were performed.The participants enrolled in the study provided written informed consent.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- RBP4 in diabetes: RBP4 in diagnosed diabetes.
  Interventions: Other: Exposure factors
- RBP4 in pre-diabetes (pre-DM): RBP4 in pre-diabetes (pre-DM).
  Interventions: Other: Exposure factors
- RBP4 in DM-CVD: RBP4 in diabetic cardiovascular disease.
  Interventions: Other: Exposure factors
- RBP4 in CVD: RBP4 in single coronary artery disease.
  Interventions: Other: Exposure factors
- RBP4 in NC: RBP4 in healthy controls.
  Interventions: Other: Exposure factors

INTERVENTIONS:
Other: Exposure factors — Exposure factors，such as diet，exercise，environment

SUMMARY:
Retinol-binding protein 4 (RBP4) may affects obesity development and the development of obesity-related diseases including insulin resistance, type 2 diabetes, steatohepatitis and cardiovascular disease. This study aims to examine the involvement of RBP4 in patients with diagnosed diabetes, diabetic cardiovascular disease, pre-diabetes (pre-DM) and healthy controls during the progression of T2DM, and to evaluate the ability of RBP4 to predict cases of diabetes with an elevated risk of cardiovascular complications . Along with animal experiment.

DETAILED DESCRIPTION:
A total of 500 Chinese patients admitted to the First Affliated Hospital of Xi'an Jiaotong University (Xi'an, China) between March 2020 and March 2022 were recruited to investigate the RBP4 profles. Peripheral blood samples are drawn at the initial medical examination, in the morning after a fast of at least 8 h, and immediately stored at -80˚C until the sphingolipid measurements were performed.

Blood pressure, WC, hip circumference (HC), body weight and body height were measured by a trained physician. The participants enrolled in the study provided written informed consent.

ELIGIBILITY:
Inclusion Criteria:

T2DM:

* Fasting plasma glucose (FPG)≥7.0 mmol/l;
* 2 h plasma glucose (2hPG) ≥11.1 mmol/l;
* glycated hemoglobin (HbA1c) level ≥6.5%;
* random plasma glucose ≥11.1 mmol/l plus symptoms of hyperglycemia;
* T2DM diagnosed previously.

Pre-DM was defned as follows:

* FPG ≥5.6-6.9 mmol/l
* 2hPG 7.8-11.0 mmol/l
* HbA1c 5.7-6.4%.

Exclusion Criteria:

* type 1 diabetes
* liver or kidney disorders.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 500 Chinese patients admitted to the First Affliated Hospital of Xi'an Jiaotong University (Xi'an, China) between March 2020 and March 2022 were recruited to investigate the RBP4 profles. The different groups were matched for age, sex and BMI.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
serum RBP4 level | 2022.3
  serum RBP4 level in DM, pre-DM, CVD, DM-CVD and healthy controls.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Sui, doctor, Study Director — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China